CLINICAL TRIAL: NCT04627051
Title: A Prospective, Single-Centre Study Investigating the Clinical Use and Safety of the Jetstream Atherectomy With Drug Coated Balloon (Ranger) for the Treatment of Dysfunctional Arterio-Venous Graft Stenosis
Brief Title: Atherectomy and Drug Coated Balloon for the Treatment of Arterio-Venous Graft Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5673
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-11

CONDITIONS: Dysfunctional Arterial-venous Grafts
MeSH Terms: interventions — Atherectomy; Angioplasty, Balloon

STUDY DESIGN:
Intervention Model Description: Treatment of Jetstream™ atherectomy device and Ranger ™ drug coated balloons
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dysfunction AV graft (Experimental): Dysfunctional AV graft stenosis treated with atherectomy and drug coated balloon angioplasty
  Interventions: Device: Atherectomy and balloon angioplasty

INTERVENTIONS:
Device: Atherectomy and balloon angioplasty — Atherectomy and balloon angioplasty of arterial-venous graft stenosis

SUMMARY:
This single-centre, single-arm, prospective study will enroll 30 subjects presenting with clinical and hemodynamic abnormalities in arteriovenous graft (AVG) in the arm. Subjects will be treated with the Jetstream™ atherectomy device and Ranger™ Drug Coated Balloons (DCB). Subjects will be followed up clinically via office visit or phone visit at 6 and 12 months post procedure. This study is to demonstrate safety and assess the clinical use and outcomes of the Jetstream ™atherectomy device and Ranger™ DCB for the treatment of dysfunctional AV graft.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breastfeeding female ≥18 years of age;
* Subject is willing to provide informed consent, and is willing to comply with the protocol-required follow up visits;
* Target lesion must be a mature arteriovenous graft presenting with any clinical, physiological or hemodynamic abnormalities warranting angiographic imaging as defined in the K/DOQI guidelines;
* Subject has a target lesion at the venous anastomosis of the AVG;
* Successful crossing of the stenosis;
* Each lesion length is ≤20mm, which may include tandem lesions that are ≤20mm apart

Exclusion Criteria:

* Subject is currently participating in an investigational drug or device study which has not yet reached its primary endpoint or was previously enrolled into this study;
* Subject has a non-controllable allergy to contrast;
* Subject has more than 3 lesions in the access circuit requiring intervention;
* Target lesion diameter >10mm;
* A thrombosed access or an access with a thrombosis treated ≤30 days prior to the index procedure;
* Prior surgical interventions of the access site ≤30 days before the index procedure;
* Target lesion is located within a bare metal or covered stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Primary Patency (TLPP) through 6 months | within 6 months post intervention
  50% re-stenosis of the target lesion

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided